CLINICAL TRIAL: NCT05797467
Title: Adjuvant Chemotherapy Combined With Targeted Therapy Versus Adjuvant Chemotherapy Alone in the Treatment of Stage T3-4N2 Colorectal Cancer:A Multicenter, Randomized, Phase III Clinical Trail
Brief Title: Adjuvant Chemotherapy Combined With Targeted Therapy or Not in the T3-4N2 Colorectal Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, Principal Investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1010CG(2022)-03
Record Dates: First submitted 2023-03-20; First posted 2023-04-04 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Chemotherapy Effect
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combining targeted therapy group (Experimental): Adjuvant chemotherapy with targeted therapy
  Interventions: Drug: FOLFOX chemotherapy regimens; Drug: Bevacizumab
- Single adjuvant chemotherapy group (Sham Comparator): Adjuvant chemotherapy alone
  Interventions: Drug: FOLFOX chemotherapy regimens

INTERVENTIONS:
Drug: FOLFOX chemotherapy regimens — Chemotherapy regimens recommended include oxaliplatin-based CapeOx or FOLFOX regimens, or single-agent 5-FU/LV, capecitabine, or combination with targeted therapy.
  Other Names: CapeOx regimens
Drug: Bevacizumab — Targeted therapy regimens are recommended based on gene testing results. For colorectal cancer patients with KRAS/NRAS/BRAF gene mutations, it is recommended to use Bevacizumab in combination with chemotherapy. For right-sided colon cancer patients with wild-type KRAS/NRAS/BRAF genes, it is recommended to use Bevacizumab. For left-sided colon and rectal cancer patients with wild-type KRAS/NRAS/BRAF genes, it is recommended to use Cetuximab.When using targeted therapy in combination with chemotherapy, the treatment course should be synchronized with chemotherapy (Bev 5mg/kg iv d1 or Cet 500mg/m2 iv d1).
  Other Names: Cetuximab
  Arms: Combining targeted therapy group

SUMMARY:
The goal of this clinical trial] is to compare in resectable stage T3-4N2 colorectal cancer. The main question it aims to answer is: whether the use of targeted therapy in combination with adjuvant chemotherapy is associated with improved disease-free survival (DFS) compared to adjuvant chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes, aged 18-75 years;
2. Pathologically confirmed pT3-4N2 stage colorectal adenocarcinoma after surgery;
3. ASA grade < IV and/or ECOG performance status score ≤ 2 points;
4. Fully understand and voluntarily sign the informed consent form for this study.

Exclusion Criteria:

1. A history of other malignant tumors;
2. Patients with severe liver, kidney, cardio-pulmonary, coagulation dysfunction, or underlying diseases that cannot tolerate chemotherapy;
3. Patients allergic to any component in the study;
4. Patients with severe uncontrollable recurrent infections or other severe uncontrollable concurrent diseases;
5. Patients with other factors that may affect the study results or lead to premature termination of the study, such as alcoholism, drug abuse, other serious diseases requiring comprehensive treatment (including mental illness), and severe abnormalities in laboratory tests;
6. Patients with emergent surgery due to intestinal obstruction, intestinal perforation, intestinal bleeding, etc.;
7. Patients with a history of severe mental illness;
8. Pregnant or lactating women;
9. Patients with other clinical or laboratory conditions that the investigators consider inappropriate for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2030-04-01 (Estimated); Study Completion 2033-04-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years after operation.
  disease-free survival (DFS) is defined as the time from the date of surgery for colorectal cancer to the occurrence of tumor recurrence or metastasis, or death from any cause.
5-year disease-free survival | 5 years after operation.
median of disease-free survival | 5 years after operation.

SECONDARY OUTCOMES:
3-year overall survival | 3 years after recruited.
  Overall survival (OS) is defined as the time from the date of randomization to the date of death from any cause. For patients who are still alive at the time of the final analysis, the date of the last contact will be recorded.
5-year overall survival | 5 years after recruited.
Complications | 5 years after recruited.
  When evaluating the safety and tolerability of adjuvant therapy, researchers typically assess adverse events (AEs) based on their incidence and severity, and then grade them according to the NCI CTCAE version 5.0. NCI CTCAE 5.0 categorizes AEs into 5 grades based on severity, including grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), and grade 5 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliate Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided